CLINICAL TRIAL: NCT06208267
Title: The Impact of Additional Post-operative Doses of Tranexamic Acid on Pain, Mobility and Bleeding Following Total Hip and Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Tranexamic Acid Use on Pain, Mobility and Bleeding Following Total Hip and Total Knee Arthroplasty
Acronym: TXA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Anthony Albers, MD, Director of Orthopaedic Research, Orthopaedic Surgeon, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-1082
Record Dates: First submitted 2023-11-02; First posted 2024-01-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Bleeding
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be recruited in the pre-operative clinic for surgery and randomized once all paperwork is completed. This randomization will be completed by a research assistant and transmitted to pharmacy to allow for the delivery of the proper medication packet. Neither the patient nor the treating physician will be made aware of the group to which the patient has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1)Standard care: 1G TXA IV (Active Comparator): 1 gm TA IV given prior to incision and 1G TXA IV during cementation or closure
  Interventions: Drug: Tranexamic acid
- 2) Standard + 1G oral TXA - 0 and 8 hours post-operatively (Active Comparator): Standard + 1G oral TXA given at 0 and 8 hours post-operatively
  Interventions: Drug: Tranexamic acid
- 3) Standard + 1G oral TXA given at 0, 8, 16 and 24 hours post-operatively (Active Comparator): Standard + 1G oral TXA given at 0, 8, 16 and 24 hours post-operatively
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — This is a 3 arm RCT using the three dosage regimens mentioned above. Placebo doses will be provided for the 0, 8, 16 and 24 hours without TXA
  Other Names: CYKLOKAPRON

SUMMARY:
Tranexamic acid (TXA) is an anti-fibrinolytic agent developed in the 1960s that has been safely used to reduce blood loss, transfusion rates and bleeding-associated mortality in trauma, obstetrics and orthopedic surgery, including hip fracture care and arthroplasty.

The efficacy and safety profile of TXA has been extensively studied in numerous clinical trials and observational studies. Its wide range of applications, combined with its favourable risk-benefit ratio, has led to the incorporation of TXA into clinical guidelines and protocols worldwide.

This RCT aims to compare the current standard dosing for TXA to additional TXA doses given orally post-operatively for THA and TKA patients. The goal is to compare the following between study groups: visible bleeding on post-operative dressing, mobilization (steps, amount of time moving around), pain (visual analog scale), function (Oxford hip and knee scales) and ROM at four to six weeks.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) and total hip arthroplasty (THA) are some of the most common surgical procedures performed in elderly patients, with the main indication being end-stage osteoarthritis. While these procedures can result in a significant amount of bleeding, pain and stiffness post-operatively, they have been increasingly performed as day surgeries and with reduced length of stay.

Tranexamic acid (TXA) is an anti-fibrinolytic agent developed in the 1960s that has been safely used to reduce blood loss, transfusion rates and bleeding-associated mortality in trauma, obstetrics and orthopedic surgery, including hip fracture care and arthroplasty.

The efficacy and safety profile of TXA has been extensively studied in numerous clinical trials and observational studies. Its wide range of applications, combined with its favourable risk-benefit ratio, has led to the incorporation of TXA into clinical guidelines and protocols worldwide.

The current standard of care at St-Mary's for TXA use is one gram given intravenously (IV) at the beginning of the replacement and one gram given during cementation. However, despite the established benefits of TXA, the optimal dosing regimen continues to be an area of ongoing research and discussion.

TXA and post-operative hemoglobin and hematocrit levels The use of TXA in knee and hip arthroplasty has been shown to have clear and significant benefits in reducing the post-operative drop in hemoglobin (Hb) and hematocrit (Hct) but the duration of use has ranged from a single pre-operative dose to a prolonged 14-day course. Researchers reported higher post-operative Hb and Hct following THA and TKA using a three-day course of TXA compared to a single pre-operative dose of 1.5g. However another study, showed no added benefit of the addition of a second post-operative dose to the single pre-operative dose. Similarly, an randomized controlled trial (RCT) comparing TXA doses at pre, during and three hours post-operative to the same with additional doses at six and 12 hours and showed no added benefit of the additional two doses on Hb or Hct levels. In contrast to this, three RCTs performed in 2019 and 2021 showed improved Hb and Hct levels with TXA use beyond a minimum of seven hours post-operatively and two involved the use of TXA given by mouth (PO), which is ideal in the ambulatory setting.

TXA and Ambulation/Motion The majority of the studies involving varying doses of TXA following THA and TKA have not assessed articular motion nor ambulation post-operatively. These can have an impact on patient satisfaction as well as the ability to mobilize and be able to leave the hospital earlier. TXA was compared to placebo and demonstrated that patients who received TXA ambulated 20% more during physiotherapy sessions. Several TXA regimens with patients receiving a minimum of three post-operative doses (maximum of four post-operative doses were studied),showed having significantly better range of motion (ROM) than patients who received less. Additionally, these patients reported less post-operative pain.

TXA and Complications

No increase in adverse events were reported in any of these studies following prolonged TXA use. Cardiovascular events, deep vein thrombosis (DVT), pulmonary embolism (PE), renal failure or superficial thrombosis were not different among study groups in the rare cases where they occurred, even with oral TXA given for up to 14 days post-operatively

. At St-Mary's Hospital, we perform a large number of TKAs and THAs, around 1100 per year (600 knees, 500 hips), making us the most productive hospital performing these procedures in Québec. Also, partly driven by the constraints of the pandemic over the past three years, we have successfully and safely reduced the length of stay for our patients and converted hundreds of patients to day surgery. Bleeding, however, remains a significant source of patient anxiety, with 10% of our ambulatory cases needing additional CLSC care or even return to hospital. Rapid mobilization and decrease in post- operative pain are also key factors for a rapid and safe discharge from hospital.

In this RCT, we aim to compare our current standard dosing for TXA to additional TXA doses given orally post-operatively for our THA and TKA patients. We will be the first of this type of study to assess patient mobility using a wearable device that will allow for precise measurement of step counts, amount of time moving around and sleep times. Also new compared to previous studies, will be our assessment of bleeding complications requiring intervention and needs for additional hospital or nursing visits, both of which have and impact on the cost of care. Pain (VAS scale), function (Oxford hip and knee scales) and ROM will also be assessed at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

° All adults undergoing primary TKA and THA at St-Mary's Hospital

Exclusion Criteria:

* Age < 18 years
* Known hypersensitivity or allergy to TXA
* Previous history of thromboembolic disease
* Active malignancy (all current cancers other than local skin cancer)
* Significant renal disease (hematuria, dialysis, kidney transplant)
* History of convulsions
* Known defective colour vision
* Inability or unwillingness to use MyMobility app
* Unable to communicate in French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Step counts at 24 and 48 hours post -operative | Post-operative
  We hypothesize that patients receiving additional doses of TXA will mobilize more at 24 and 48 hours post- operatively and that this will be dose-dependent.

SECONDARY OUTCOMES:
Range of motion (ROM) of the hip (if applicable): | 4 - 6 weeks post op
  Measuring ROM of the hip taken pre-operatively, post-operatively and 4 to 6 weeks post-operatively if patient received a total hip arthroplasty (THA)
Range of motion (ROM) of the knee (if applicable): | 4 - 6 weeks post op
  Measuring ROM of the knee taken pre-operatively, post-operatively and 4 to 6 weeks post-operatively if patient received a total knee arthroplasty (TKA).
Patient self-assessment of functionality and pain measured pre-operatively, 4 to 6 weeks postoperatively, 3 months postoperatively and 6 months post-operatively following total hip arthroplasty utilizing the Oxford Hip Score (OHS): | 4 to 6 weeks postoperatively, 3 months postoperatively and 6 months post-operatively
  Minimal value of 0 and maximal value of 48. The higher scores indicate more satisfactory joint function.
Patient self-assessment of functionality and pain measured pre-operatively, 4 to 6 weeks postoperatively, 3 months postoperatively and 6 months post-operatively following total knee arthroplasty utilizing the Oxford Knee Score (OKS): | 4 to 6 weeks postoperatively, 3 months postoperatively and 6 months post-operatively
  joint function.
Bleeding Complications requiring intervention | Return to the emergency room or bleeding complications will be noted.
  Bleeding that require a specific intervntion from CLSC/Clinic/Hospital visits
Daily step counts | Post-operative day 0,1,2,3,5,7 and 4 to 6 weeks postoperatively.
  To be measured with an application (MyMobility) on a smartphone or smartwatch used by the patient. This is a numerical value simply describing the number of steps taken by the patient on a day-to-day basis. This measurement will be collected pre-operatively (until OR), on post-operative day 0,1,2,3,5,7 and 4 to 6 weeks postoperatively.
Measure of quality of life using the 12-Item Short Form Survey (SF-12): | This measurement will be taken pre-operatively, 4 to 6 weeks postoperatively, 3 months postoperatively and 6 months post-operatively.
  Regarding minimum and maximum values, there are two summary scores that are reported from the SF-12: there is a mental component score (MCS-12) and a physical component score (PCS-12). The scores may also be reported as Z-scores where a difference would be compared to the population average.
  In the literature, SF-12 results have also been computed as a range going from a minimum value of 0 to a maximum value of 100, where higher scores indicate better physical and mental health functioning.
Assessment and screening for depression and anxiety in patients utilizing the Hospital Anxiety Depression Scale (HADS) : | Pre-operative
  Minimum score of 0 and maximum score of 21. The higher scores indicate higher distress.
Reported pain self-reported in patient journal and possibly in-patient charts: | These journals and/or in-patient charts will be verified on postoperative day 0,1,2,3,5 and 7.
  This is a numerical value. Patient journals and/or in-patient charts, if applicable, would be screened for frequency of opioid use as a way of evaluating pain management post-operatively.
Assessment of catastrophic thinking related to pain utilizing the Pain Catastrophizing Scale (PCS): | Pre-operative
  Minimum score of 0 and maximum score of 52. The higher scores indicate higher levels of catastrophizing.
Reported pain using the visual analog pain (VAS) scale: | This measurement will be collected on postoperative day 0, 1,2,3,5 and 7.
  The pain VAS scale involves a numerical rating scale or a descriptive rating scale that progressively goes from a minimal value indicating severe pain to a maximal value indicating good pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mutch, MDCM, FRCSC, Principal Investigator — St. Mary's Hospital Centre
Locations (1):
- St. Mary's Hospital Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No